CLINICAL TRIAL: NCT01645241
Title: Evolutive Potential of Embryos Obtained From Oocytes After Luteal Phase Ovarian Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Collaborators: FUNDACION DEXEUS SALUT DE LA DONA (Unknown); Ayudas Merck Serono de Investigación 2012 (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEX005
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2013-03

CONDITIONS: INFERTILITY; Fertility Preservation; Ovulation Induction; Vitrification; Oocyte Donation
Keywords: Ovarian stimulation; Luteal phase; Egg donors; Fertility preservation
MeSH Terms: conditions — Infertility | interventions — Gonadotropins; Ovulation Induction; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lutheal phase ovarian stimulation (Experimental): Early luteal phase Controlled ovarian hyperstimulation: we will administer in the 13th-15th cycle day simultaneously 0.25 mg/day of ganirelix to induce luteolysis and FSHr (dose according to BMI and AFC )IU/day for controlled ovarian hyperstimulation until achieving criteria for hCG , to induce final oocyte maturation. Mature oocytes will be vitrified. After warming, oocytes will be inseminated by ICSI with the recipients partners semen sample . Recipient endometrium will be primed with estrogen and progesterone , and embryo transfer will be performed on the 3rd day 3 of embryo cleavage.
  Interventions: Drug: gonadotropins plus GnRH antagonists; Drug: ganirelix

INTERVENTIONS:
Drug: gonadotropins plus GnRH antagonists
  Other Names: Ovarian stimulation
Drug: ganirelix
  Other Names: the investigators will administer in the 13th-15th cycle day simultaneously 0.25 mg/day of ganirelix

SUMMARY:
The purpose of this study is to evaluate the clinical pregnancy rate per embryo transfer in oocytes recipients obtained after ovarian stimulation during the luteal phase of oocytes donors . This study will be performed in egg recipients and donors but this type of treatment is meant to be implemented in fertility preservation patients

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women, 18-35 years old, FSH levels < 10 mIU/ml; AFC> 10
* regular cycles
* BMI < 28
* signed informed consent

Recipients:

* Infertile women eligible for oocytes donation
* BMI < 35
* Signed informed consent form

Exclusion Criteria:

-Polycystic ovarian syndrome, gonadotropins allergy

Recipients:

* Women eligible for oocytes donation
* BMI >35
* Uncontrolled Endocrine Pathology

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | six weeks after transfer procedure

SECONDARY OUTCOMES:
Number of Mature oocytes | Day of oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Martínez, PhD, Principal Investigator — Fundación Dexeus Salut de la Dona
Locations (1):
- Departamento de Obstetricia Ginecologia y Reproducción. Institut Universitari Dexeus, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Sonmezer M, Turkcuoglu I, Coskun U, Oktay K. Random-start controlled ovarian hyperstimulation for emergency fertility preservation in letrozole cycles. Fertil Steril. 2011 May;95(6):2125.e9-11. doi: 10.1016/j.fertnstert.2011.01.030. Epub 2011 Feb 3. PMID 21292255
- [Background] von Wolff M, Thaler CJ, Frambach T, Zeeb C, Lawrenz B, Popovici RM, Strowitzki T. Ovarian stimulation to cryopreserve fertilized oocytes in cancer patients can be started in the luteal phase. Fertil Steril. 2009 Oct;92(4):1360-1365. doi: 10.1016/j.fertnstert.2008.08.011. Epub 2008 Oct 18. PMID 18930226
- [Derived] Martinez F, Clua E, Devesa M, Rodriguez I, Arroyo G, Gonzalez C, Sole M, Tur R, Coroleu B, Barri PN. Comparison of starting ovarian stimulation on day 2 versus day 15 of the menstrual cycle in the same oocyte donor and pregnancy rates among the corresponding recipients of vitrified oocytes. Fertil Steril. 2014 Nov;102(5):1307-11. doi: 10.1016/j.fertnstert.2014.07.741. Epub 2014 Aug 22. PMID 25154677
- See also: Related Info — http://www.dexeus.com